CLINICAL TRIAL: NCT05852041
Title: A Pilot Study of rhPSMA-PET MRI Imaging for the Detection of Clinically Actionable Prostate Cancer Among Men Who Are Otherwise Candidates for Active Surveillance
Brief Title: rhPSMA-73 PET-MRI Imaging for the Detection of Prostate Cancer Among Men Who Are Otherwise Candidates for Active Surveillance
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ashley Ross MD, PhD, Associate Professor, Department of Urology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NU 22U05; NCI-2023-02187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00218970; NU 22U05 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Masking Description: A read will completed for the PET portion of the examination by a nuclear medicine trained radiologist who is blinded to the mpMRI portion of the exam.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rhPSMA, PET-MRI, mpMRI) (Experimental): Patients receive rhPSMA-7.3 IV then undergo PET-MRI and mpMRI of the prostate on study. Patients also undergo Decipher test at screening and MRI-PET prostate biopsy or radical prostatectomy within 90 days per standard of care.
  Interventions: Procedure: Biopsy of Prostate; Genetic: Decipher Prostate Cancer Test; Other: Flotufolastat F-18 Gallium; Procedure: Magnetic Resonance Imaging; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Radical Prostatectomy

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo MRI/PET prostate biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Genetic: Decipher Prostate Cancer Test — Undergo decipher
  Other Names: Decipher; Decipher Metastasis Test; Decipher Test
Other: Flotufolastat F-18 Gallium — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; rhPSMA-7.3 (18F)
Procedure: Magnetic Resonance Imaging — Undergo PET-MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Procedure: Positron Emission Tomography — Undergo PET-MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This clinical trial evaluates whether positron emission tomography-magnetic resonance imaging (PET-MRI) using the radioactive drug radiohybrid prostate-specific membrane antigen (rhPSMA)-7.3 may help in detecting higher grade or stage disease in men with low and favorable intermediate risk prostate cancer who are candidates for active surveillance. A PET scan is a test that uses a radioactive drug and a computer to create images of how organs and tissues in the body are functioning. The radioactive drug used in this study, rhPSMA-7.3, attaches to the abnormal cells in the body at a different rate than normal cells which allows the scanner to create a detailed picture of how the body is working. An MRI scan uses strong magnets and computers to create detailed images of the soft tissue in your body. A multiparametric (mp)MRI is a type of MRI scan that creates a more detailed picture of the prostate gland. Using rhPSMA-73 with PET-MRI and mpMRI may be more effective in detecting higher grade or stage disease in men with low and favorable intermediate risk prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Measure the rate of rhPSMA-7.3-PET-MRI identified Gleason Grade Group (GG) 3-5 disease on pathology or locally advanced disease. A threshold rate of 15% detection will be considered clinically significant.

SEONDARY OBJECTIVE:

I. Assessment of safety.

EXPLORATORY OBJECTIVES:

I. Determine the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for rhPSMA-PET-MRI to detect prostate cancer in the prostate stratified by Gleason Grade Groups.

II. Correlate PET MRI findings with surgical specimens for those men who undergo surgical treatment (including assessment of pathological stage).

III. Define whether gene expression of PSMA (FOLH1) as defined on the Decipher messenger ribonucleic acid (mRNA) expression platform relates to signal intensity on PSMA scan.

IV. Determine whether Decipher genomic classifier scores, luminal / basal scores or androgen receptor activity scores relate to signal intensity on PSMA scans.

OUTLINE:

Patients receive rhPSMA-7.3 intravenously (IV) then undergo PET-MRI and mpMRI of the prostate on study. Patients also undergo Decipher test at screening and MRI-PET prostate biopsy or radical prostatectomy within 90 days per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men (Eastern Cooperative Oncology Group [ECOG] 0-1), >= 18 years old with at least 10 year life expectancy
* Histologically proven Gleason Grade Group 1 or 2 adenocarcinoma of the prostate
* Last prostate cancer containing biopsy performed within 3-15 months (mo.) prior to screening. Biopsy must have been >= 10 core biopsy and informed by prior mpMRI
* Prostate cancer categorized as low risk or favorable risk by National Comprehensive Cancer Network (NCCN) criteria (low risk is defined as T1c-T2a, prostate-specific antigen [PSA] < 10ng/ml, Gleason Grade Group 1 [Gleason 3+3=6] disease) and favorable intermediate risk as having no more than one of the following intermediate risk features, clinical T2b-T2c disease, PSA 10-20ng/ml, Gleason Grade Group 2 [Gleason score 3+4=7])
* Decipher genomic classifier score from prior biopsy >= 0.45
* Institutional Review Board (IRB)-/Independent Ethics Committee (IEC)-approved written informed consent and privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures
* Concurrent diseases and malignancies are permitted
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on the study
* Willing to undergo prostate biopsy prior to non-surgical treatment of prostate cancer and within 90 days of PET-MRI imaging

Exclusion Criteria:

* Prior radiotherapy, surgery, chemotherapy, or hormonal therapy for prostate cancer
* NCCN very low risk category (T1c and Gleason Grade Group 1 [Gleason score 3+3=6], PSA < 10 ng/mL, fewer than 3 prostate biopsy cores positive, =< 50% cancer in any core, PSA density < 0.15 ng/mL/g)
* Decipher score < 0.45
* Prior bladder outlet procedure (i.e,. holmium laser enucleation of the prostate [HoLEP], transurethral resection of the prostate [TURP], Urolift, Rezum)
* Prohibited medications: use of 5 alpha reductase inhibitor or androgen deprivation therapy (i.e., leuprolide, relugolix) within 1 month of screening
* Contra-indication or relative contra-indication to MRI (i.e., pacemaker)
* History of hip replacement
* Subject has received investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2035-06-07 (Estimated)

PRIMARY OUTCOMES:
Radio-pathological correlation between positron emession tomography-magnetic resonance imaging (PET-MRI) and prostate biopsy or radical prostatectomy | Up to 90 days
  Will report agreement between pathology and imaging and ability of radiohybrid prostate-specific membrane antigen-7-PET-MRI to identify higher grade and stage disease as a raw percentage.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | Within 24 hours of radio-tracer injection
  Occurrence of severe adverse events occurring following imaging will be reported as a percentage. Will use the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Ross, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Jang JW, Abrams A, Jawahar A, Savas H, Yang XJ, Mehta V, Schnauss M, Schaeffer EM, Alam R, Ross AE. Detection of MRI-Invisible Disease Using PSMA PET/CT in a Patient Considering Focal Therapy. Case Rep Urol. 2025 Mar 26;2025:2981515. doi: 10.1155/criu/2981515. eCollection 2025. PMID 40177325